CLINICAL TRIAL: NCT03032835
Title: Partners Calciphylaxis Biobank and Patient Registry
Brief Title: Partners Calciphylaxis Biobank
Acronym: PCB
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sagar U. Nigwekar, MD, MMSc, Assistant in Medicine, Massachusetts General Hospital
Other Study IDs: 2016P002690
Record Dates: First submitted 2017-01-23; First posted 2017-01-26 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Calciphylaxis; Calcific Uremic Arteriolopathy; End Stage Renal Disease; Chronic Kidney Diseases
Keywords: Calciphylaxis; Warfarin; Dialysis
MeSH Terms: conditions — Calciphylaxis; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Plasma, serum, DNA and tissue samples (e.g. skin)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: No intervention

SUMMARY:
Calciphylaxis, a vascular calcification disorder, is a rare and serious disorder characterized by calcification of dermal arterioles.

There are significant gaps in the understanding of the pathophysiology and risk factors for calciphylaxis. At present, there is no effective treatment. Uncertain pathobiology, rare incidence and lack of collaborative approach have been some of the major limiting factors towards treating calciphylaxis.

The Partners Calciphylaxis Biorepository (PCB) aims to address these gaps within calciphylaxis research by utilizing existing and, when necessary, developing new infrastructure to support the consent of patients and the collection of dedicated samples for a calciphylaxis repository.

DETAILED DESCRIPTION:
Calciphylaxis, a vascular calcification disorder, is a rare and serious disorder characterized by calcification of dermal arterioles.

There are significant gaps in the understanding of the pathophysiology and risk factors for calciphylaxis. At present, there is no effective treatment. Uncertain pathobiology, rare incidence and lack of collaborative approach have been some of the major limiting factors towards treating calciphylaxis.

The Partners Calciphylaxis Biorepository (PCB) aims to address these gaps within calciphylaxis research by utilizing existing and, when necessary, developing new infrastructure to support the consent of patients and the collection of dedicated samples for a calciphylaxis repository.

This repository is working in collaboration with the Partners Biobank as they will still be receiving samples from the PCB and storing them and distributing them according to their own procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old
2. Skin lesions consistent with calciphylaxis diagnosis as determined by the treating clinician
3. Informed of the investigational nature of the study and sign written Informed consent OR are eligible for surrogate consent process based on impaired decision making

Exclusion Criteria:

1. Patients <18 years of age
2. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with skin lesions consistent with calciphylaxis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improvement in calciphylaxis skin lesions | 6 months
  Skin lesions will be assessed by investigators at baseline (entry into study) and at 6 months to determine whether there is improvement. The investigators will determine clinical, laboratory and genetic predictors of this outcome in calciphylaxis patients.

SECONDARY OUTCOMES:
Number of patients with >30% improvement in pain severity | 4weeks
  Pain severity will be assessed by investigators at baseline (entry into study) and at 4 weeks to determine whether there is improvement. Pain is measured using Wong-Baker Faces pain rating scale. The investigators will examine clinical, laboratory and genetic predictors of this outcome in calciphylaxis patients.
Time to death in patients with calciphylaxis | Up to 5 years
  Time to death is defined as time from the diagnosis of calciphylaxis to death (or to the end of follow up). The investigators will examine clinical, laboratory and genetic predictors of this outcome in calciphylaxis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar U Nigwekar, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nigwekar SU, Bloch DB, Nazarian RM, Vermeer C, Booth SL, Xu D, Thadhani RI, Malhotra R. Vitamin K-Dependent Carboxylation of Matrix Gla Protein Influences the Risk of Calciphylaxis. J Am Soc Nephrol. 2017 Jun;28(6):1717-1722. doi: 10.1681/ASN.2016060651. Epub 2017 Jan 3. PMID 28049648
- [Background] Nigwekar SU, Zhao S, Wenger J, Hymes JL, Maddux FW, Thadhani RI, Chan KE. A Nationally Representative Study of Calcific Uremic Arteriolopathy Risk Factors. J Am Soc Nephrol. 2016 Nov;27(11):3421-3429. doi: 10.1681/ASN.2015091065. Epub 2016 Apr 14. PMID 27080977
- [Background] Nigwekar SU, Kroshinsky D, Nazarian RM, Goverman J, Malhotra R, Jackson VA, Kamdar MM, Steele DJ, Thadhani RI. Calciphylaxis: risk factors, diagnosis, and treatment. Am J Kidney Dis. 2015 Jul;66(1):133-46. doi: 10.1053/j.ajkd.2015.01.034. Epub 2015 May 7. PMID 25960299
- [Derived] Wen W, Krinsky S, Kroshinsky D, Durant O, He J, Seethapathy R, Hillien SAS, Mengesha B, Malhotra R, Chitalia V, Nazarian RM, Goverman J, Lyons KS, Nigwekar SU. Patient-Reported and Clinical Outcomes Among Patients With Calciphylaxis. Mayo Clin Proc Innov Qual Outcomes. 2023 Jan 24;7(1):81-92. doi: 10.1016/j.mayocpiqo.2022.12.006. eCollection 2023 Feb. PMID 36712824
- See also: Link to publications — https://www.ncbi.nlm.nih.gov/pubmed?term=((Nigwekar)%20AND%20((Calciphylaxis)%20OR%20(Calcific%20uremic%20arteriolopathy)))